CLINICAL TRIAL: NCT03472378
Title: Effects of DFN-15 on Migraine With Allodynia
Brief Title: Can DFN-15 Terminate Migraine With Allodynia?
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Rami Burstein, PhD, Beth Israel Deaconess Medical Center (Unknown); Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Principal Investigator, Brian Grosberg, Brian M Grosberg, MD, Hartford Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HHC-2017-0224
Record Dates: First submitted 2018-02-20; First posted 2018-03-21 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Migraine With Aura; Migraine Without Aura; Allodynia
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura; Hyperalgesia | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Treatment Group (Experimental): DFN-15
  Interventions: Drug: DFN-15
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DFN-15 — Oral Solution of 4.8 mL containing 120 mg of DFN-15
  Other Names: Celecoxib
  Arms: Active Treatment Group
Other: Placebo — Oral Solution of 4.8 mL containing 0 mg of DFN-15
  Arms: Placebo Group

SUMMARY:
The majority of migraineurs seeking secondary or tertiary medical care develop cutaneous allodynia during the course of migraine, a sensory abnormality mediated by sensitization of central trigeminovascular neurons in the spinal trigeminal nucleus. Triptan therapy can render allodynic migraineurs pain-free within a narrow window of time (20-120 min) that opens with the onset of pain and closes with the establishment of central sensitization. This calls for the development of drugs that can tackle ongoing central sensitization and render allodynic migraineurs pain-free after the window for triptan therapy has expired. There are two main objectives the investigators seek to achieve from this study: to determine whether oral administration of DFN-15 (solution of a COX2 inhibitor, Celecoxib) terminates migraine attacks when given to allodynic participants 3 hours after attack onset; and to determine whether mechanical and heat allodynia that develop during acute migraine attacks could be reversed by late (> 3hrs after attack onset) treatment with DFN-15. Participants will be recruited from the Headache Center and randomized in a double-blinded fashion to receive either the active drug (DFN-15) or placebo in a ratio of 4:1.The participants will be instructed to return to the clinic during a migraine. At the 'during-migraine' visit, which will begin 3 hours after onset of headache, the investigators will document headache intensity, associated symptoms, and mechanical and heat pain threshold (first) before treatment (at 180 min after onset of headache) and (second) at a 120 min after treatment (5 hours after headache onset). Based on our prior experience studying migraine patients, the investigators plan to screen 100 patients to achieve 50 participants completing the 2 study visits as planned. The active drug group will consist of 80/100 patients and 20/100 patients will receive the placebo. The study will be terminated as soon as the first 40 participants who received the DFN-15 and first 10 patients who received placebo completed visit 2.

ELIGIBILITY:
Inclusion Criteria:

* History of migraine with or without aura for at least 3 years, based on the International Classification of Headache disorders
* Two or more migraine attacks per month on average during the year prior to enrollment
* Ability to give written consent to enrollment

Exclusion Criteria:

* Fifteen or more headache days per month, on average
* Aspirin or NSAID induced asthma or allergy
* Sulfa allergy
* Any woman who is pregnant or lactacting
* History of any of the following: Coronary artery bypass surgery, heart attack, angina, stroke, serious gastrointestinal bleeding, peptic ulcer disease, and/or chronic kidney disease
* Medical Conditions requiring the use of diuretics or daily anticoagulants
* Severe uncontrolled medical problems or medications that may influence measurements

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Headache Pain Intensity | Up to 6 months
  The proportion of patients demonstrating a decrease in their headache pain intensity is greater than 50% (post-treatment compared to pre-treatment). Pain intensity will be measured with a visual analog scale from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Allodynia | Up to 6 months
  The proportion of patients demonstrating allodynia before and after treatment; allodynia to thermal stimuli is defined as pain threshold < 41 degrees Celsius, and to mechanical stimuli as pressure pain threshold of < 30 g.

CONTACTS AND LOCATIONS:
Locations (1):
- Hartford HealthCare Headache Center, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT03472378/Prot_SAP_000.pdf